CLINICAL TRIAL: NCT00504946
Title: The Effect of Glucocorticosteroid and Vitamin D3 Administration and Montelukast Treatment on Early Clinical and Immunological Effect of Allergen-Specific Immunotherapy in Asthmatic Children, Double-Blind, Placebo-Controlled Study
Brief Title: Pharmacological Modulations of Allergen-Specific Immunotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Medical Universtity of Lodz, Department of Pediatrics and Allergy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN-168-05-KE
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Asthma
Keywords: allergen immunotherapy premedication
MeSH Terms: conditions — Asthma | interventions — Prednisone; Lactose; Budesonide; Cholecalciferol; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- I (Active Comparator)
  Interventions: Drug: prednisone, lactose
- II (Active Comparator)
  Interventions: Drug: prednisone, colecalciferol, lactose
- III (Placebo Comparator)
  Interventions: Drug: lactose
- A (Active Comparator)
  Interventions: Drug: montelukast sodium
- B (Placebo Comparator)
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: prednisone, lactose — Allergen immunotherapy (build-up phase)premedication with orally administrated in the day of immunotherapy:
  20mg prednisone+ 0.3mg lactose
  Other Names: Miflonide; Pulmicort
  Arms: I
Drug: prednisone, colecalciferol, lactose — Allergen immunotherapy (build-up phase)premedication with orally administrated in the day of immunotherapy:
  20mg prednisone + 1000j colecalciferol + 0.3mg lactose
  Other Names: Miflonide; Pulmicort
  Arms: II
Drug: lactose — Allergen immunotherapy (build-up phase)premedication with orally administrated in the day of immunotherapy:
  0.3mg lactose
  Other Names: Miflonide; Pulmicort
  Arms: III
Drug: montelukast sodium — Allergen immunotherapy (build-up phase)premedication with montelukast sodium. Children 6-14 years received 5 mg of montelukast and children > 14 years old received 10mg oral tablet once daily at bedtime
  Other Names: Miflonide; Pulmicort
  Arms: A
Drug: lactose — Allergen immunotherapy (build-up phase)premedication with 0,3mg lactose once daily at bedtime
  Other Names: Miflonide; Pulmicort
  Arms: B

SUMMARY:
There is mounting evidence that successful allergen immunotherapy (SIT) functions through the induction of different subset of Treg including Foxp3 positive cells, therefore additional strategies to enhance this property are highly attractive. Based on previous findings we assumed that combine allergen immunotherapy with non-specific treatments such as glucocorticosteroids and vitamin D3 as well as montelukast sodium treatment might enhanced allergen tolerance induction and improved clinical effectiveness of allergen-specific immunotherapy

DETAILED DESCRIPTION:
There is mounting evidence that successful allergen immunotherapy (SIT) functions through the induction of different subset of Treg including Foxp3 positive cells, therefore additional strategies to enhance this property are highly attractive. Since corticosteroids directly induce the development of an IL-10-synthesizing regulatory T-cell population (Tr1) and this effect can be greatly increased with vitamin D3 treatment we , we assumed that combine allergen immunotherapy with non-specific treatments such as glucocorticosteroids and vitamin D3 as well as montelukast sodium treatment might enhanced allergen tolerance induction and improved clinical effectiveness of allergen-specific immunotherapy, therefore we conducted the stud comparing the effect of glucocorticosteroid, glucocorticosteroid with vitamin D3 or montelukast sodium on early immunological and clinical effect of allergen-specific immunotherapy in asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

* allergic asthma with regular symptoms requiring long-term treatment with inhaled corticosteroids
* disease duration of at least 2 years
* sensitisation only to house dust mites
* resting FEV1 of more or equal 70%

Exclusion Criteria:

* sensitization to allergens other than house dust mites
* discontinuation of SIT from any reasons
* need of a daily dose below 200 or above 800 mcg of budesonide or equivalent
* other chronic disease including vitamin D3 deficiency and/or resistance which could influence the results of the study or the patient's ability to participate in the study as judged by the investigator
* medications that resulted in patient exclusion included: inhaled long acting β2-agonist, leukotriene modifiers, β-blockers (eye drops included) or oral corticosteroids within 6 month before the pre-study visit.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Regulatory T cell (CD4+CD25+Foxp3 positive) induction measured in peripheral blood mononuclear cells | First visit, second visit (after 3 months) and third visit (after 12 months of immunotherapy)

SECONDARY OUTCOMES:
Cytokine (IL-10, TGF-beta1, IL-4, IL-5, IL-13) determination in supernatants from peripheral blood mononuclear cells culture. | First visit, second visit (after 3 months) and third visit (after 12 months of immunotherapy)
diary card evaluation with asthma free days estimation, lung function measurement and analysis of reduction of the inhaled corticosteroids dose | Visit first and third visit (after 12 months of immunotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Majak, MD, PhD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD, PhD, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz Lodz, Poland, Lodz, Poland